CLINICAL TRIAL: NCT00724633
Title: Effect of Lowering the Dialysate Sodium on Blood Pressure in Hemodialysis Patients: a Randomized Controlled Trial.
Brief Title: Effect of Lowering the Dialysate Sodium on Blood Pressure in Hemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-08-252; 15153
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Hemodialysis
Keywords: dialysate; sodium; hemodialysis; blood pressure; thirst; intradialytic symptoms; interdialytic weight gain; extracellular fluid balance; mechanisms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Other): standard dialysate Na 140 mEq/L
  Interventions: Other: Lowering the dialysate sodium
- 2 (Active Comparator): dialysate sodium equal to patient's predialysis serum Na
  Interventions: Other: Lowering the dialysate sodium
- 3 (Active Comparator): dialysate sodium lower than patient's predialysis plasma sodium
  Interventions: Other: Lowering the dialysate sodium

INTERVENTIONS:
Other: Lowering the dialysate sodium — Please see above

SUMMARY:
Patients currently receiving hemodialysis will be randomized to receive 1 of 3 dialysate sodium prescriptions. The effects on blood pressure, interdialytic weight gain, thirst, and intradialytic symptoms will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients on 3 times weekly hemodialysis of at least 3 months
* elevated average ambulatory blood pressures
* current dialysate sodium prescription 140mEq/L
* average pre-dialysis serum sodium <140mEq/L

Exclusion Criteria:

* frequent intradialytic hypotension
* estimated life expectancy <1 year
* non-adherence to dialysis prescription
* pregnancy
* inability or unwillingness to complete study measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Ambulatory blood pressure | 3 months
  Ambulatory blood pressure to be taken over 24 hours at 4 week intervals throughout the study

SECONDARY OUTCOMES:
thirst | 3 months
QOL Scores (KDQOL, mins to recovery) | 3 months
intradialytic hypotension rate, intradialytic symptoms | 3 months
mechanistic outcomes: interdialytic weight gain, extracellular fluid water, sodium ionic mass balance | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rita Suri, MD, MSc, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Center, London, Ontario, Canada

REFERENCES:
- [Derived] Marshall MR, Wang MY, Vandal AC, Dunlop JL. Low dialysate sodium levels for chronic haemodialysis. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD011204. doi: 10.1002/14651858.CD011204.pub3. PMID 39498822